CLINICAL TRIAL: NCT01904669
Title: Prospective Evaluation of the Elements of Pregnancy Study
Brief Title: Internet-based Study of Fertility and Early Pregnancy (PEEPS)
Acronym: PEEPS
Status: Completed | Type: Observational
Sponsor: Courtney D.Lynch, PhD MPH (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Courtney D.Lynch, PhD MPH, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012H0128; 1R03HD073504-01 (NIH)
Record Dates: First submitted 2013-07-15; First posted 2013-07-22 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Fertility; Infertility; Pregnancy; Abortion, Spontaneous
Keywords: Fertility; Infertility; Pregnancy; Conception; Behavioral; Lifestyle; Preconception Care; Women's Health; Abortion, Spontaneous; Cohort Studies; Epidemiology; Internet
MeSH Terms: conditions — Infertility; Abortion, Spontaneous; Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women who are trying to conceive: Women ages 18-44 without a history of fertility problems who are in a stable relationship with a male partner who have regular access to the Internet and have been trying to conceive <3 months.

SUMMARY:
The purpose of this study is to assess the feasibility of conducting an Internet-based prospective pregnancy study with preconception enrollment with women completing daily journals for up to 12 months while trying to conceive and weekly through pregnancy if it occurs.

DETAILED DESCRIPTION:
There is a dearth of knowledge regarding the role that preconception health plays in fertility and early pregnancy loss. Classical methods of conducting prospective pregnancy studies with preconception enrollment to answer these questions are time-consuming in terms of recruitment efforts and expensive to carry out. The purpose of this project is to assess the feasibility of conducting an Internet-based prospective pregnancy study with preconception enrollment in the United States using the gold standard data collection approach of daily diaries during the trying to conceive period. We will accomplish this by enrolling 200 females of reproductive age who attempting to conceive and following them for up to 12 months and through pregnancy for those who become pregnant. Feasibility will be assessed by measuring: the number of women who screen eligible, the number of women who enroll, and compliance with journal use over time. We will also estimate the incidence of infertility, pregnancy and pregnancy loss as well as compare the demographics of women who enroll to the demographics of women who participate in community-based prospective pregnancy studies with preconception enrollment. The data from this project will be used to assess the feasibility of launching a larger prospective pregnancy study that is appropriately powered to examine the impact of preconceptional lifestyle factors on the incidence of infertility and early pregnancy loss.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Ages 18-44
* In a stable relationship
* Sexually active with a male partner
* Reliable daily access to the Internet

Exclusion Criteria:

* Woman or her partner has a known fertility problem
* Trying to conceive for three or more months.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We are looking for women ages 18-44 who are planning a pregnancy and have been trying to conceive for <3 months. Women must have reliable daily access to the Internet. The woman and her male partner may not have any known fertility problems.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Number enrolled | One year

SECONDARY OUTCOMES:
Completeness of data collection | Following 9-21 months of data collection
  Percentage of the study that the participant completed: baseline questionnaire (Y/N); daily trying to conceive journals (%); weekly pregnancy journals (%); and delivery information (%).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Medicine, Columbus, Ohio, United States

REFERENCES:
- See also: PEEPS website — https://peeps.osumc.edu